CLINICAL TRIAL: NCT01186705
Title: A Phase II Clinical And Translational Study Of MK-2206 In Patients With Metastatic KRAS-Wild-Type, PIK3CA-Mutated, Colorectal Cancer
Brief Title: Clinical And Translational Study Of MK-2206 In Patients With Metastatic KRAS-Wild-Type, PIK3CA-Mutated, Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-068
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Results first posted 2015-04-21 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: MK-2206; colon; rectal; 10-068
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MK-2206 (Experimental): This will be a single-arm, phase II study of the AKT inhibitor MK-2206 in patients with KRAS-wild-type, PIK3CA-mutated, colorectal cancer whose tumors have progressed through standard chemotherapy regimens.
  Interventions: Drug: MK-2206

INTERVENTIONS:
Drug: MK-2206 — Patients will receive MK-2206 orally in a once weekly dose of 200mg. There will be no dose escalation. Patients will be treated until disease progression or unacceptable side effects.

SUMMARY:
The purpose of this study is to test a new drug called MK-2206 for metastatic colorectal cancer. This drug is being tested in a subgroup of patients with colorectal cancer whose tumors have changes in certain genes that may make them more likely to respond to this new medication. As tumors develop, the cells within the tumor acquire mutations within genes, allowing them to grow more effectively. We will be testing your tumor for mutations involving two genes - KRAS and PIK3CA. Patients whose tumors have a normal copy of the KRAS gene and a mutation within the PIK3CA gene will be eligible to participate in this study.

This study is a phase 2 study. The goal of a phase 2 study is to find out what effects, good and/or bad, a new treatment has against a certain type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have metastatic colorectal cancer that has been histologically or cytologically-confirmed at MSKCC and has failed to respond to appropriate standard therapy regimens. There is no limit on the number of prior treatment regimens permitted.
* Patient is male or female and ≥18 years of age on the day of signing informed consent.
* Patient must have performance status of 0 or 1 on the ECOG Performance Scale.
* Patient must have adequate organ function as indicated by the following laboratory values:
* Absolute neutrophil count (ANC) ≥1,500 /μL
* Platelets ≥100,000 /μL
* Hemoglobin ≥9 g/dL
* Serum creatinine or calculated creatinine clearance ≤1.5 x upper limit of normal (ULN) OR ≥60 mL/min for patients with creatinine levels >1.5 x institutional ULN
* Serum total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 x ULN
* AST (SGOT) and ALT (SGPT) ≤3 x ULN or ≤5 x ULN in patients with known liver metastasis
* Prothrombin time (PT)/INR ≤1.5 x ULN
* Partial thromboplastin time (PTT)≤1.5 x ULN
* Fasting serum glucose ≤120 mg/dl
* HBA1C ≤8%
* Potassium in normal range
* The patient has a tumor that has wild type KRAS (absence of mutations at codons 12 or 13), and mutant PIK3CA (presence of mutations in exons 20 or 9).
* Female patient of childbearing potential who are not surgically sterilized must have a negative serum or urine pregnancy test β-hCG within 72 hours prior to receiving the first dose of study medication.
* Patient, or the patient's legal representative, has voluntarily agreed to participate by giving written informed consent.
* Patient is able to swallow capsules and has no surgical or anatomical condition that will preclude the patient from swallowing and absorbing oral medications on an ongoing basis.

Exclusion Criteria:

* Patient who has had chemotherapy, radiotherapy, or biological therapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C), or who has not recovered from the adverse events due to previous agents administered more than 4 weeks prior to Study Day 1. If the patient has residual toxicity from prior treatment, toxicity must be ≤ Grade 1.
* Patients must be at least 4 weeks post major surgical procedure, and all surgical wounds must be fully healed.
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of Study Day 1.
* Patient has known CNS metastases and/or carcinomatous meningitis.
* Patient has a primary central nervous system tumor.
* Patient has known hypersensitivity to the components of study drug or its analogs.
* Patient has a history or current evidence of clinically significant heart disease including:
* Clinically significant congestive heart failure, unstable angina pectoris,
* Clinically significant cardiac arrhythmia,
* History or current evidence of a myocardial infarction during the last 6 months, and/or a current ECG tracing that is abnormal in the opinion of the treating Investigator,
* QTc prolongation ≥450 msec (Bazett's Formula), Patient with evidence of clinically significant bradycardia (HR <50), or a history of clinically significant bradyarrhythmias such as sick sinus syndrome, 2nd degree AV block (Mobitz Type 2).
* Patient with uncontrolled hypertension (i.e., > 160/90 mHg SiBP). Patients who are controlled on antihypertensive medication will be allowed to enter the study.
* Patient at significant risk for hypokalemia (e.g., patients on high dose diuretics, or with recurrent diarrhea)
* Patient with poorly controlled diabetes (HBA1C >8%)
* Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Patient is, at the time of signing informed consent, a regular user (including -recreational use‖) of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
* Patient is breastfeeding or expecting to conceive or father children within the projected duration of the study.
* Patient is known to be Human Immunodeficiency Virus (HIV)-positive
* Patient has known history of Hepatitis B or C or active Hepatitis A.
* Patient has symptomatic ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions is eligible.
* Patient is receiving treatment with oral corticosteroids (note: inhaled corticosteroids are permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saltz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-2206
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MK-2206
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate (ORR)
Description: in patients with metastatic colorectal cancer with known PIK3CA mutations and wild type KRAS, to single agent MK-2206. Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | MK-2206
Number analyzed (Participants) | 1
participants
  Progression of Disease | 1
  Stable Disease | 0

ADVERSE EVENTS:
Arm/Group | MK-2206
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2206 (N=1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
White blood cell descreased (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes